CLINICAL TRIAL: NCT04781127
Title: An Open Label Home-administered Transcranial Direct Current Stimulation (tDCS) Clinical Trial of Unipolar Depression
Brief Title: Home-administered tDCS for Treatment of Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMI-F10
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Unipolar Depression; Treatment Resistant Depression
Keywords: tDCS
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Active tDCS (Experimental): Active Transcranial Direct Current Stimulation (tDCS), Soterix Medical mini-CT tDCS stimulator
  Interventions: Device: Soterix Medical mini-CT tDCS stimulator

INTERVENTIONS:
Device: Soterix Medical mini-CT tDCS stimulator — Stimulation will last 30 minutes per day, 5 days per week, for 5 weeks, then 3 days per week for 1 week and then 1 day per week for 4 weeks.
  Other Names: Soterix Medical ElectraRx; Soterix Medical SNAPpad

SUMMARY:
This study will determine the safety and efficacy of home administered tDCS in adults with unipolar depression. The device used to administer tDCS will be the Soterix Medical 1X1 mini-CT. 32 tDCS sessions of 30 minutes each will be delivered over 10 weeks.

DETAILED DESCRIPTION:
The Soterix Medical 1X1 mini-CT will be used to determine the safety and efficacy of home-based transcranial direct current stimulation (tDCS) in treating unipolar depression. Specifically efficacy will be determined by change in MADRS score from baseline to the 10 week follow-up. Feasibility and compliance will be determined by low drop out rate and percentage of scheduled sessions completed. Self-reported mood scores will be evaluated using the Quick Inventory of Depressive Symptomatology (QIDS-SR) and Quality of Life enjoyment and Satisfaction Questionnaire Form (Q-LES-Q-SF). All visits will be performed via telephone or video conference. Subjects will be taught to operate the tDCS system and complete a tolerability check. The treatment course will consist of an acute phase of 28 tDCS sessions conducted Monday - Friday over 6 weeks. This is followed by a taper of 4 tDCS sessions spaced 1 week apart. Patients who meet criteria for clinical response (>=50% improvement in MADRS) may continue with maintenance treatments of once a week for 2 months and once every 2 weeks for the remaining 3 months. Mood assessments will be conducted at baseline, 2 weeks, 4 weeks and 6 weeks in the acute treatment phase. In the taper phase, assessments wil be conducted at 1 month (end of taper), 3 and 6 months following completion of the acute phase. All assessments in the acute treatment phase and the taper phase will have a +/- 1 week collection window.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients that meet criteria for diagnosis of MDD according to DSM-V-TR and confirmed with the Mini International Neuropsychiatric interview.
* Currently experiencing a major depressive episode of at least 4 week's duration as part of a unipolar depression
* Scored at least 20 on the MADRS at trial entry
* Patient's antidepressant medication is stable for at least 30 days prior to MADRS screening
* Female patients are allowed if not pregnant and are using a medically acceptable method of contraception, if of childbearing potential

Exclusion Criteria:

* DSM-V-TR psychotic disorder
* Drug or alcohol abuse or dependence in the preceding 3 months
* Concurrent benzodiazepine medication
* High suicide risk
* History of clinically defined neurological disorder or insult
* Metal in the cranium or skull defects
* Subjects with an implanted pump, neurostimulator, cardiac pacemaker or defibrillator
* Skin lesions on scalp at the proposed electrode sites
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Mood | Baseline, at the end of Weeks 2, 4 ,6 during the acute phase, at completion of taper phase (end of Week 10) and during the Follow-up period (end of Weeks 18 and 30)
  Mood will be assessed with the Montgomery Asberg Depression Rating Scale (MADRS). Patients who meet criteria for clinical response (>=50% improvement in MADRS) may continue with maintenance treatments of once a week for 2 months and once every 2 weeks for the remaining 3 months.

SECONDARY OUTCOMES:
Self-Reported Mood Score | Weeks 1-10. Patients who receive maintenance sessions will also report before sessions 33-46 (Weeks 11-30)
  Patients will enter daily mood scores before each treatment session on a scale of 0-10 (0= feeling normal and not depressed at all and 10= feeling as depressed as possible) on the web interface.
Quick Inventory of Depressive Symptomology (QIDS-SR) | Weeks 1-10. Patients who receive maintenance sessions will also report at the end of Weeks 11-18, 20, 22, 24, 26, 28, 30
  Patients will enter responses at the end of each week on the web interface. (16 question survey with higher score for more severe symptoms)
Quality of Life Enjoyment and Satisfaction Questionnaire Form (Q-LES-Q-SF) | Weeks 1-10. Patients who receive maintenance sessions will also report at the end of Weeks 11-18, 20, 22, 24, 26, 28, 30
  Patients will enter responses at the end of each week on the web interface. (16 question survey with answers between 1-5 where higher score represents better outcomes)
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, at the end of Weeks 2, 4 ,6 during the acute phase, at completion of taper phase (end of Week 10) and during the Follow-up period (end of Weeks 18 and 30)
  Patients will respond to questions about suicidal ideation and behavior, where "yes" or "no" answers indicate level of risk (low, moderate or high). More "yes" answers indicate worse outcomes.
Self-report Columbia Suicide Severity Rating Scale (C-SSRS) | Weeks 1-10
  Patients will enter scores before each treatment session on the web interface about suicidal ideation and behavior, where "yes" or "no" answers indicate level of risk (low, moderate or high). More "yes" answers indicate worse outcomes.
Adverse Effects: Pain | Weeks 1-10
  Participants will enter any side effects experienced, their severity (mild, moderate, severe), pain scores based on the Wong-Baker pain scale and temporal relationship with the tDCS session (before, during, after).
Adverse Effects: Suicidal Ideation | Weeks 1-10
  Participants will enter a score using item 9 of the Beck Depression Inventory (range from 0 = "I don't have any thoughts of killing myself." to 3 = "I would kill myself if I had the chance.")

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Datta, PhD, Principal Investigator — Soterix Medical Inc.
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Moffa AH, Sampaio-Junior B, Borrione L, Moreno ML, Fernandes RA, Veronezi BP, Nogueira BS, Aparicio LVM, Razza LB, Chamorro R, Tort LC, Fraguas R, Lotufo PA, Gattaz WF, Fregni F, Bensenor IM; ELECT-TDCS Investigators. Trial of Electrical Direct-Current Therapy versus Escitalopram for Depression. N Engl J Med. 2017 Jun 29;376(26):2523-2533. doi: 10.1056/NEJMoa1612999. PMID 28657871